CLINICAL TRIAL: NCT02497898
Title: A Randomized Controlled Clinical Trial of Cytokine-induced Killer (CIK) Cells Treatment in Patients With Refractory Non-Hodgkin Lymphoma
Brief Title: Treatment of CIK for Patients With Refractory Non-Hodgkin Lymphoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First People's Hospital of Changzhou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RNHL001
Record Dates: First submitted 2015-06-29; First posted 2015-07-15 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-06

CONDITIONS: Lymphoma, Non-Hodgkin
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- regular chemotherapy (No Intervention): Patients after chemotherapy are just followed up.
- CIK regimen (Experimental): Patients after chemotherapy will receive at least 3 cycles of Cytokine-induced killer cells (CIK) treatment every 3 months.
  Interventions: Biological: Cytokine-induced killer cells (CIK)

INTERVENTIONS:
Biological: Cytokine-induced killer cells (CIK) — Cytokine-induced killer (CIK) cells are able to eradicate lymphomas and other malignancies. CIK cells are generated by incubation of peripheral blood lymphocytes with an anti-cluster of differentiation 3 (anti-CD3) monoclonal antibody, interleukin-2 (IL-2), interleukin-1 (IL-1) and interferon-gamma.
  Arms: CIK regimen

SUMMARY:
The purpose of this study is to study the safety and efficacy of chemotherapy usage followed by CIK transfusion in refractory and/or chemoresistant lymphomas.

DETAILED DESCRIPTION:
Autologous cytokine-induced killer (CIK) cells transfusion(>2*10^9 cells count) within 2 weeks after regular chemotherapy every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed as non-Hodgkin lymphoma with negative effect of regular chemotherapy, and need further therapy

Exclusion Criteria:

* patients refuse the therapy or have no tolerance for the therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2015-07; Primary Completion 2038-07 (Estimated); Study Completion 2040-07 (Estimated)

PRIMARY OUTCOMES:
Progression-Free-Survival (PFS) | 1 month

SECONDARY OUTCOMES:
Overall Survival (OS) | 1 month

OTHER OUTCOMES:
Lactic Dehydrogenase (LDH) | 1 month